CLINICAL TRIAL: NCT03460340
Title: Randomized Sham-controlled Study of Deep Transcranial Magnetic Stimulation (dTMS) as a Treatment for Patients With Fibromyalgia
Brief Title: dTMS as a Treatment for Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHA-17-18
Record Dates: First submitted 2018-02-04; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Studying Efficacy of dTMS in FM
Keywords: dTMS; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: randomized control trial (RCT)
Who Masked: Participant
Masking Description: participants do not know if they are getting the DTMS treatment or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FM group (Experimental): patients diagnosed with Fibromyalgia receiving dTMS treatment.
  Interventions: Device: prefrontal deep rTMS of H1 Coil
- placebo group (Sham Comparator): patients diagnosed with Fibromyalgia receiving sham- treatment.
  Interventions: Device: prefrontal deep rTMS of H1 Coil

INTERVENTIONS:
Device: prefrontal deep rTMS of H1 Coil — prefrontal deep rTMS of H1 Coil

SUMMARY:
Purpose: The purpose of the study is to explore the efficacy of H1 deep TMS for the treatment of FMS.

Design: Prospective randomized sham controlled trial Study Population & sample size:forty (40) FMS subjects between 18-80 years of age.

No. of Centers: Four centers-

1. Shalvata Mental Health Center, Tel -Aviv University, Israel.
2. Soraski medical center, Tel-Aviv University, Israel.
3. Sheba Medical Center, Tel-Aviv University, Israel
4. Beer-Yakov Mental Health Center, Tel-Aviv University, Israel. Duration and intensity of Treatment: All subjects will receive prefrontal deep rTMS of H1 Coil (75 trains of 2 seconds, 20 Hz, with 20 seconds inter-train intervals, up to 120% of motor threshold, a total of 3000 pulses per session), for 4 weeks, 5 days a week, overall 20 sessions.

Name of device: The Brainsway Ltd. H1-Coil

Study Endpoints: Clinical outcome:

primary outcome Change in self-reported average pain intensity over the last 24 hours will be measured at the end point with the numerical scale (0 = no pain, 10 = maximal pain imaginable) of the VAS-FIQ.

secondary outcome

1. Change of sensory and affective pain dimensions will be measured at the end point using the McGill Pain Questionnaire.
2. Change of the impact of pain and FMS on quality of life, will be measured at the end point using the BPI items for pain interference.
3. change of sensitivity to painful stimuli will be evaluated by physical measurements:

   * WPI
   * SSS
4. Changes in cognitive functions in domains of attention, working memory, spatial memory, executive functions and social cognition will be measured at the beginning and end point of the study using the Penn Web-Based Computerized Neurocognitive Battery (WebCNP).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years.
* Patients who continue to take their administered medications or patients who stopped ineffective administered medications
* Concomitant medication for pain and sleep disorders will be allowed provided the dose administered had been stable for at least 2 weeks before enrollment and remains stable throughout the study.
* Gave informed consent for participation in the study.

Exclusion Criteria:

* Subjects will be excluded if evidence is found of inflammatory rheumatic disease, autoimmune disease, or other painful disorders that might confound assessment of FMS pain.
* Subjects diagnosed with a current primary (Axis I) psychiatric condition according to Diagnostic and Statistical Manual of Mental Disorders-IV criteria, including anxiety disorders, not including major depression or major personality disorder. Subject with a history of substance abuse and pregnant women will be excluded as well.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of head injury.
* History of seizure or heat convulsion.
* History of epilepsy or seizure in first degree relatives.
* History of frequent or severe headaches.
* Use of hearing aids for hearing loss.
* Known history of cochlear implants.
* History of drug abuse or alcoholism during the last year.
* Serious and unstable medical condition, which is likely to exacerbate or endanger the patient during the treatment period.
* Significant difficulties in language or communication.
* Subjects declared as legally incompetent, with an appointed physical guardian and/or cannot sign informed consent due to cognitive incompetence.
* Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
change in self-reported average pain intensity over the last 24 hours | at the beginning of each session, before stimulation (Subjects will undergo 5 courses per week for 4 weeks)
  self-reported average pain intensity over the last 24 hours will be measured with numerical scale (0 = no pain, 10 = maximal pain imaginable) of the VAS-FIQ- self-reported average pain intensity scale

SECONDARY OUTCOMES:
Change of sensory and affective pain dimensions | at baseline, once a week during trial period (4 weeks), and at follow-up visit (2 weeks after the end of the treatments)
  Change of sensory and affective pain dimensions -using the McGill Pain Questionnaire (16 items rated between 0 "not at all" - 3 "very strong")
Change of the impact of pain and FMS on quality of life | at baseline, once a week during trial period (4 weeks), and at follow-up visit (2 weeks after the end of the treatments)
  Change of the impact of pain and FMS on quality of life- using the BPI- items rated between 1 "functioning as usual" to 10 "very affected by the pain")
Changes in cognitive functions in domains of attention, working memory, spatial memory, executive functions and social cognition | baseline and end point (after 4 weeks)
  Changes in cognitive functions in domains of attention, working memory, spatial memory, executive functions and social cognition - using the the Penn Web-Based Computerized Neurocognitive Battery (WebCNP).

IPD SHARING:
Plan to Share IPD: Undecided
no IPD planned to be shared at this moment